CLINICAL TRIAL: NCT05024877
Title: The Efficacy and Safety of Hetrombopag for Low/Intermediate-1 Risk MDS With Thrombocytopenia
Brief Title: Hetrombopag for Low/Intermediate-1 Risk MDS With Thrombocytopenia
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Bing Han, Docter, Peking Union Medical College Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HBP-MDS-001
Record Dates: First submitted 2021-08-19; First posted 2021-08-27 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2021-09

CONDITIONS: MDS
MeSH Terms: interventions — hetrombopag; Stanozolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hetrombopag treatment group (Experimental): stanozolol 2mg tid + Hetrombopag (started with 5mg/day and increased by 2.5mg/day every 2 weeks if the platelet count remains less than 20×10e9/L and reduced if the platelet count reaches over than 150×10e9/L, the maximum dosage is 15mg/day)
  Interventions: Drug: Hetrombopag; Drug: Stanozolol Tablets

INTERVENTIONS:
Drug: Hetrombopag — Hetrombopag would be given started with 5mg/day and increased by 2.5mg/day every 2 weeks if the platelet count remains less than 20×10e9/L and reduced if the platelet count reaches over than 150×10e9/L, the maximum dosage is 15mg/day)
Drug: Stanozolol Tablets — Stanozolol would be given 2mg tid.

SUMMARY:
Myelodysplastic syndrome (MDS) is a kind of clonal myeloid tumor. The major manifestation is decrease of tri-lineages of blood due to ineffective and abnormal hematopoiesis, some of which can progress to acute myeloid leukemia. According to the international prognosis scoring system (IPSS) of MDS, about 10% low/intermediate risk-1 MDS patients have severe thrombocytopenia (PLT < 30 × 109/ L). These patients have both decreased platelet count and platelet dysfunction, resulting in a high risk of bleeding. In the new prognostic score, such as IPSS-r, the degree of thrombocytopenia is regarded as a poor prognostic factor. Platelet transfusion is mainly used in the treatment of this kind of patients. The indications of transfusion include bleeding events or severe platelet count reduction (< 10 × 109 / L). However, platelet transfusion can only lead to short-term platelet elevation, while repeated transfusion increases the possibility of infection and ineffective platelet transfusion. TPO is a newly discovered hematopoietic promoting factor, which can specifically bind to the TPO receptor on the cell and participate in the regulation of proliferation, differentiation, maturation and division of megakaryocyte to form functional platelet. The efficacy and safety of the TPO receptor agonists eltrombopag and romiplostim in the treatment of thrombocytopenia in low/intermediate risk-1 MDS patients have been successfully confirmed in foreign studies. Hetrombopag is a new kind of a TPO receptor agonists which is highly specific platelet stimulating factor. At present, there is no large report on the application of Hetrombopag in such patients. The purpose of this study is to explore the short-term and long-term therapeutic effect and safety of Hetrombopag on low/intermediate risk-1 MDS patients.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed MDS, IPSS low / intermediate risk-1
2. In the 4 weeks before inclusion, the average value of platelets was ≤ 30 × 10e9 / L, or < 50 × 10e9 / L with bleeding events
3. Patients with EPO due to anemia and G-CSF due to severe neutropenia can be included, and the dosage will not change during trial
4. ECOG 0-2 points
5. Able to sign informed consent

Exclusion Criteria:

1. Pregnant or lactating
2. IPSS intermediate risk-2 / high risk MDS
3. More than 5% of myeloblasts in bone marrow
4. Myelofibrosis
5. Previous transplantation or ATG treatment within 6 months
6. Previous use of TPO or other TPO receptor agonists
7. Active infection or tumor
8. Thromboembolic or hemorrhagic disease
9. Serious heart disease, including unstable angina, congestive heart failure, arrhythmia, 1-year history of myocardial infarction
10. Baseline liver and kidney function: ALT / ASL over than 3 times normal upper limit, TBIL over than 2 times normal upper limit, and creatinine over than 2 times normal upper limit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
overall response rate at 6 months | 6 month
  Overall Response Rate (ORR) Defined as the Number of Participants Who Met the Criteria of Either Complete Response (CR) or Partial Response (PR) at 6 months

SECONDARY OUTCOMES:
percentage of side effects at 12 months | 12 months
  percentage of side effects would be recorded during the study and be calculated according to CTCAE 5.0 at 12 months
ISTH-BAT (ISTH bleeding assessment tool) | 12 months
  to evaluate the severity of bleeding, the proposed normal cutoffs are >=4 in adult males, >=6 in adult females, and >=3 in children, respectively
change of platelet transfusion | 12 months
  the total amount of platelet transfusion per month
onset time for overall response | through study completion, an average of 1 year
  onset time for complete and partial response
duration of overall response | through study completion, an average of 1 year
  during time for complete and partial response
life quality for MDS patients | 12 months
  life quality for MDS patients by QoL-E questionaire（scores range from 0 to 100，higher scores mean better).
the change of myeloblasts in bone marrow and peripheral blood | 12 months
  the increased number of myeloblasts in bone marrow and peripheral blood
incidence of progression to high-risk MDS or leukemia | 12 months
  incidence of progression to high-risk MDS or leukemia

CONTACTS AND LOCATIONS:
Overall Officials: Bing Han, Docter, Study Director — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
protocol, consent form, clinical data would be available by personal contact
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 10 years
Access Criteria: personal contact including emails

REFERENCES:
- [Background] Mei H, Liu X, Li Y, Zhou H, Feng Y, Gao G, Cheng P, Huang R, Yang L, Hu J, Hou M, Yao Y, Liu L, Wang Y, Wu D, Zhang L, Zheng C, Shen X, Hu Q, Liu J, Jin J, Luo J, Zeng Y, Gao S, Zhang X, Zhou X, Shi Q, Xia R, Xie X, Jiang Z, Gao L, Bai Y, Li Y, Xiong J, Li R, Zou J, Niu T, Yang R, Hu Y. A multicenter, randomized phase III trial of hetrombopag: a novel thrombopoietin receptor agonist for the treatment of immune thrombocytopenia. J Hematol Oncol. 2021 Feb 25;14(1):37. doi: 10.1186/s13045-021-01047-9. PMID 33632264